CLINICAL TRIAL: NCT05554887
Title: Effect of Thoracic Manipulation on Muscle Strength and Pressure Pain Threshold in Healthy Individuals With Rhomboid Latent Trigger Point: A Randomized Sham Controlled Study.
Brief Title: Effect of Thoracic Manipulation on Latent Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Şule ŞİMŞEK, Principal investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.07.2022/11
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Trigger Points
Keywords: latent trigger point; thorasic manipulation; muscle strength; pressure pain threshold

STUDY DESIGN:
Intervention Model Description: randomised sham controlled study involving 2 parallel groups
Who Masked: Outcomes Assessor
Masking Description: All these evaluations will be carried out by a blind evaluator who does not know which group the participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrust manipulation Group (Experimental): Participants undergoing thrust manipulation
  Interventions: Other: Thrust manipulation
- Sham thrust manipulation group (Sham Comparator): Participants undergoing sham thrust manipulation
  Interventions: Other: Sham thrust manipulation

INTERVENTIONS:
Other: Thrust manipulation — Participants will be positioned prone and the clinician will perform a high-speed, low-amplitude thrust into the most symptomatic segment of the thoracic spine. TM type, thrust direction, and number of thrusts will be at the clinician's discretion and will be based on the individualized assessment of the patient.
  Arms: Thrust manipulation Group
Other: Sham thrust manipulation — The same protocol will be applied as the push thoracic manipulation application, but no push will be applied.
  Arms: Sham thrust manipulation group

SUMMARY:
The aim of this study is to investigate the effect of one session thoracic manipulation on pressure pain threshold and rhomboid muscle strength in healthy individuals with latent trigger point.

DETAILED DESCRIPTION:
Within the scope of the study, all individuals studying at Sarayköy Vocational School and volunteering to participate in the study will be screened.Immediately after determining the latent trigger points in the rhomboid muscles, the participants will be randomized by computer method and divided into 2 groups. Participants who underwent thrust thoracic manipulation will form the study group, and participants who received sham thrust thoracic manipulation will form the control group.Pressure pain threshold will be evaluated with an algometer and rhomboid muscle strength will be evaluated with a hand dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* not having any systemic disease
* not having any neuromuscular deficit
* To be defined as inactive (less than 30 minutes of moderate physical activity five times a week) according to the minimum activity guidelines published by the American College of Sports Medicine

Exclusion Criteria:

* Being actively involved in any sport
* Participating in a regular exercise program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | up to 3 months
  assessed with algometer
rhomboid muscle strength | up to 3 months
  assessed with hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Şule Şimşek, Phd, Study Director — Phd faculty member
Locations (1):
- Şule Şimşek, Denizli, Sarayköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanney WJ, Puentedura EJ, Kolber MJ, Liu X, Pabian PS, Cheatham SW. The immediate effects of manual stretching and cervicothoracic junction manipulation on cervical range of motion and upper trapezius pressure pain thresholds. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):1005-1013. doi: 10.3233/BMR-169573. PMID 28505955
- [Background] The effect of lower cervical and upper thoracic spinal manipulative therapy on pressure algometer readings of rhomboid and infraspinatus muscles by influencing the fascial tension of the spiral line: Doctoral dissertation, Johannesburg: University of Johannesburg, 2015.